CLINICAL TRIAL: NCT02027233
Title: Efficiency in Population of Influenza Vaccination for Flu Prevention of the Hospitalized Adults
Brief Title: Clinical Trial to Assess the Influenza Vaccination of the Hospitalized Adults
Acronym: FLUVAC EV-03
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: C13-47; 2013-A01204-41 (Registry Identifier: IDRCB)
Record Dates: First submitted 2013-12-12; First posted 2014-01-06 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Severe Acute Respiratory Infection
Keywords: Prevention; Influenza and others respiratory viruses; Adults hospitalized; Vaccines; Effectiveness, surveillance
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nasopharyngeal sample (Experimental): Rapid completion of nasopharyngeal within 24 hours after hospitalization without exceeding 7 days after the onset
  Interventions: Other: nasopharyngeal sample

INTERVENTIONS:
Other: nasopharyngeal sample — The nasopharyngeal sample will be used to find the types and subtypes of influenza virus and other respiratory viruses (VRS, SARS-CoV-2 and others).

SUMMARY:
This study assesses the seasonal of influenza vaccine effectiveness in adults hospitalised with laboratory-confirmed influenza through a network of hospitals in France.

Also, To better understand the burden of other respiratory viruses such as respiratory syncytial virus (RSV) and SARS-CoV-2 in hospitalized adults, we need to describe and quantify the population hospitalized due to theses other respiratory viruses.

DETAILED DESCRIPTION:
Influenza vaccination strategies aim at protecting high-risk population from severe outcomes. Estimating the effectiveness of seasonal vaccines against influenza related hospitalisation is important to guide these strategies. The main objective is to measure the population effectiveness of influenza vaccine in patients hospitalized with virologically confirmed influenza laboratory result during all influenza seasons from 2013/2014 to 2021/2022 in a French hospital network. An interim analysis is provided for each influenza season and a global analysis of all seasons.

Each year, we also collect data from other respiratory viruses such as respiratory syncytial virus (RSV) on the hospitalized population. The data for three years confirm that, although RSV is less common than influenza in patients with flu-like symptom (4% of 1452 patients), it is responsible for serious complications at a higher frequency than influenza, especially in the elderly and immunosuppressed patients. To better understand the burden of disease of RSV infection in hospitalized adults, we need to start patients recruitment sooner at the start of the VRS epidemic.

With the recent emergence of the COVID-19 pandemic and our participation in European projects within the framework of COVID-19 surveillance, the FLUVAC study is an opportunity to collect additional data in patients hospitalized with a severe acute respiratory illness (SARI) which may be due to respiratory infection with an influenza virus or other respiratory viruses including SARS-CoV-2. We therefore propose to collect clinical (chronic diseases, comorbidities, intensive care), epidemiological and virological data throughout the year in adult patients hospitalized for suspected CO-VID-19.

This is a study "case-control" involving a nasopharyngeal sample for all hospitalised patients presenting a SARI within seven days. Cases will be patients RT-PCR positive for influenza. Controls will be patients negative for any influenza virus.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year
* Affiliated with social security health insurance
* Written informed consent
* Patients hospitalized for at least 24 hours for one of the reasons indicated in Table 1 of protocol
* Presence of Influenza-like syndrome before the hospitalization (even if symptoms are not present at the time of inclusion), or less than 48 hours after the hospitalization
* Rapid completion of nasopharyngeal sample after hospitalization without exceeding 7 days after the onset of Influenza-like syndrome

Exclusion Criteria:

* Realization of nasopharyngeal sampling more than 7 days after the onset of symptoms
* Contraindication for influenza vaccine (Hypersensitivity to the active substances, to any of the excipients and to trace eg eggs, including ovalbumin, chicken protein)
* Patients institutionalized without regular community interaction
* Previously tested positive for any influenza virus in the current season (RT-PCR, multiplex RT-PCR)
* Patient under curatorship or under guardianship whose sample was obtained as part of their medical care but not complying with the conditions of Article L1121-8 of the Code de la Santé Publique.
* Patient under curatorship or under guardianship whose sample was not obtained as part of their medical care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6173 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Measure of vaccine efficacy in population by comparing the number of influenza cases virologically documented in hospitalized patients vaccinated and unvaccinated. | 9 years
  The effectiveness of the vaccine in population will be calculated according to the formula VE = 1 - OR. an interval exact confidence of 95% will be calculated on the point estimate.

SECONDARY OUTCOMES:
Measure of vaccine efficacy in population by age group | 9 years
  Measure of vaccine efficacy by comparing the number of influenza cases virologically documented in hospitalized patients vaccinated and unvaccinated according to age groups
Measure of vaccine efficacy in population by influenza type/subtype | 9 years
  The objective is to compare the number of influenza cases virologically documented in hospitalized patients vaccinated and unvaccinated depending on the subtypes.
Description of the population hospitalized for syndrome acute respiratory infection (SARI) | 9 years
  The objective is to :
  * Describe and quantify the influenza hospitalized population and its complications (socio-demographic, risk factors, pattern and duration of hospitalization),
  * Describe and quantify the population hospitalized due to other respiratory viruses (VRS, SARS-CoV-2).

CONTACTS AND LOCATIONS:
Overall Officials: Odile Launay, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Institut National de la Santé Et de la Recherche Médicale, Paris, France

IPD SHARING:
Plan to Share IPD: No